CLINICAL TRIAL: NCT01278472
Title: Cosmesis and Body Image After Single Port Laparoscopic or Conventional Laparoscopic Cholecystectomy: A Double Blinded Randomised Controlled Trial
Brief Title: Cosmesis and Body Image After Single Port or 4-Port Laparoscopic Cholecystectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Zurich (Other)
Responsible Party: PD Dr. med. Stefan Breitenstein, University Hospital Zurich, Division of Visceral and Transplantation Surgery
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2010-0321/4
Record Dates: First submitted 2011-01-14; First posted 2011-01-17 (Estimated); Last update posted 2011-01-17 (Estimated); Status verified 2011-01

CONDITIONS: Symptomatic Gallstone Disease
Keywords: cholecystectomy; laparoscopic; single-port; gallstones
MeSH Terms: conditions — Gallstones

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Single Port Cholecystectomy (Experimental): Laparoscopic Cholecystectomy with single port transumbilical access
  Interventions: Device: Single Port Cholecystectomy
- 4 Port Cholecystectomy (Active Comparator): Laparoscopic Cholecystectomy using 4 separate conventional trocars
  Interventions: Device: 4 Port Cholecystectomy

INTERVENTIONS:
Device: Single Port Cholecystectomy — Using transumbilical single port device: SILS Port
  Other Names: SILS PT5, Covidien Inc.
  Arms: Single Port Cholecystectomy
Device: 4 Port Cholecystectomy — using 4 separate skin incisions and 2 5mm and 2 12 mm conventional ports
  Arms: 4 Port Cholecystectomy

SUMMARY:
Laparoscopic Cholecystectomy (LC) is the treatment of choice for symptomatic gallstone disease. Single-port access cholecystectomy (SL) has been recently introduced using only one, trans-umbilical placed port. The method has been denominated as ''scarless.'' However, it is unknown whether SL significantly improves body and cosmesis images as well as the quality of life (QoL), reported directly by the patients. Furthermore SL promises to reduce postoperative pain and to be cost-effective due a faster postoperative recovery.

The aim of this Double Blind Randomized Controlled Trial (RCT) is to demonstrate whether SL is superior to LC in improving patients', body and cosmesis images as well as QoL and to analyse cost-efficiency.

Based on the sample size calculations, a total of 110 patients will be randomised to either LC or SL. The primary endpoint will be the cosmetic score. Costs, pain, time to convalescence, quality of life and complications and will also be compared as secondary endpoints.

This study will provide evidence-based patient-oriented information regarding the SL procedure and its further use.

ELIGIBILITY:
Inclusion Criteria:

1. Patients above 18 years of age for elective cholecystectomy
2. Written informed consent from the subject
3. INR < 1.4, platelet count > 50'000/mcl

Exclusion Criteria:

1. Women in pregnancy
2. Contraindications on ethical grounds
3. Severe coagulopathy (platelet < 50'000/mcl, double medication on platelet antagonists (Plavix and Aspirin), INR > 1.4
4. liver cirrhosis
5. Enrolment of the investigator, his/her family members, employees and other dependent persons

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2011-01; Primary Completion 2012-06 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Cosmetic Score | 6 weeks postoperatively
  validated score where the minimum is 3 and the maximum 24 points. A higher score signifies a greater satisfaction of the physical appearance of the scar

SECONDARY OUTCOMES:
Body Image | 6 weeks postoperatively
  validated score. A higher score signifies a better body image.
Pain | up to 6 weeks postoperatively
  Visual Analogue Scale

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Breitenstein, PD, MD, Principal Investigator — University of Zurich
Locations (1):
- University Hospital Zurich, Division of Visceral and Transplantation Surgery, Zurich, Canton of Zurich, Switzerland

REFERENCES:
- [Derived] Lurje G, Raptis DA, Steinemann DC, Amygdalos I, Kambakamba P, Petrowsky H, Lesurtel M, Zehnder A, Wyss R, Clavien PA, Breitenstein S. Cosmesis and Body Image in Patients Undergoing Single-port Versus Conventional Laparoscopic Cholecystectomy: A Multicenter Double-blinded Randomized Controlled Trial (SPOCC-trial). Ann Surg. 2015 Nov;262(5):728-34; discussion 734-5. doi: 10.1097/SLA.0000000000001474. PMID 26583659
- [Derived] Steinemann DC, Raptis DA, Lurje G, Oberkofler CE, Wyss R, Zehnder A, Lesurtel M, Vonlanthen R, Clavien PA, Breitenstein S. Cosmesis and body image after single-port laparoscopic or conventional laparoscopic cholecystectomy: a multicenter double blinded randomised controlled trial (SPOCC-trial). BMC Surg. 2011 Sep 12;11:24. doi: 10.1186/1471-2482-11-24. PMID 21910897